CLINICAL TRIAL: NCT06016218
Title: Effect of Local Application of Platelet-Rich Fibrin Scaffold Loaded With Simvastatin Versus Bone Powder on Peri-Implant Bone Changes
Brief Title: Effect of Local Application of Simvastatin Versus Bone Powder on Implant Bone Changes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 260981
Record Dates: First submitted 2023-06-12; First posted 2023-08-29 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Dental Caries Extending to Pulp; Dental Implant Failed
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PRF (Placebo Comparator): PRF alone was added to extraction site prior to implant insertion
  Interventions: Drug: Simvastatin
- SIM+ PRF (Active Comparator): PRF + 1.2mg Statin powder are inserted into the extraction site before implant insertion
  Interventions: Drug: Simvastatin
- BO+ PRF (Active Comparator): PRF + Bone powder are inserted into the extraction site before implant insertion.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Comparing Simvastatin powder with PRF to Bone Powder with PRF on Peri-implant Bone

SUMMARY:
This study is conducted A- To investigate that PRF loaded with osteopromotive pharmacological drug can be a great aid in implant rehabilitation, and whether it could be a replacement for the other high price bone graft materials or not.

This will be done through:

1. Measuring bone changes around the implant by cone beam
2. Measuring change in bone density around the implants

B- Evaluate the effect of statins on osteoblasts activity and expression of various osteogenic products in vitro.

DETAILED DESCRIPTION:
Twenty four patients requiring rehabilitation by immediate implantation in an extraction socket were recruited for this study. The Patients were divided into three groups (n=8), For the first group; immediately after extraction, PRF alone was added into the extraction socket prior to implant insertion. For the second group, PRF + 1.2mg Statin powder are inserted into the extraction site before implant insertion. For the third Group; PRF + Bone powder are inserted into the extraction site before implant insertion. A conebeam CT was used to evaluate the effect on bone changes and bone density around implant sites, for every patient in all implant groups immediately after the surgery and at follow-up time. In vitro experiment: isolation of human Adipose mesenchymal stem cells (hAd-MSCs), characterization and osteogenic differentiation will be done. The cells were divided into two groups one control group and the other statin group. Osteogenic markers were measured in both groups and statistical analysis performed

ELIGIBILITY:
Inclusion Criteria:

* Badly Broken Down Tooth requiring extraction
* Medically Free
* Any other procedures or surgeries were performed 6 months earlier

Exclusion Criteria:

* patients with systemic diseases affecting bone quality or resorption
* temporomandibular joint dysfunction
* severe attrition or parafunctional habits
* patients undergoing radiotherapy or chemotherapy
* heavy smokers
* vulnerable groups like psychologically unstable patients.

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Changes in crestal peri-imlant Bone | 12 months
  Radiographic evaluation of crestal bone changes around the studied implants

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No